CLINICAL TRIAL: NCT05079334
Title: Improving Identification and Healthcare for Patients With Inherited Cancer Syndromes: Evidence-based EMR Implementation Using a Web-based Computer Platform
Brief Title: Family History and Cancer Risk Study
Acronym: FOREST
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Georgia Wiesner, Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: 201202; U01CA232829 (NIH)
Record Dates: First submitted 2021-10-01; First posted 2021-10-15 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: Neoplastic Syndromes, Hereditary; Comparative Effectiveness Research
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators from Vanderbilt University Medical Center (VUMC), Duke University, and Meharry Medical College (MMC) are collaborating on a family health history study to deploy a family health history (FHH) platform, MeTree. Recruited participants will complete surveys, the MeTree questionnaire, and MeTree will determine the participant's cancer risk based on current guidelines. The study team will offer genetic counseling to high-risk participants. Investigators will track participant outcomes and behaviors from the use of MeTree to determine the efficiency of the use of MeTree compared to completion of pedigrees in clinic.

DETAILED DESCRIPTION:
From the earliest recognition of cancer-prone families over 100 years ago, clinicians have depended on the family health history (FHH) to identify and treat patients and family members who may have a cancer family syndrome. Once identified, patients can be offered lifesaving, evidence-based management strategies for many of these conditions. To fully realize the benefits of genetic healthcare, however, at risk individuals must be recognized, offered genetic counseling and testing, and then referred for specialized therapy or enhanced screening. While this is a promising time for these patients and families, there are significant challenges to implement a modern and efficient care delivery model across the many patients, provider, and health system stakeholders.

The practice of genetic medicine is changing as genetic discoveries are translated into new tests for an increasing number of health indications. In fact, the prevalence of high-risk individuals who are at risk for hereditary cancer has been rising due to new testing strategies. This has placed enormous pressure on the hospitals and clinics providing care for high-risk patients. Coupled with the healthcare systems need for greater efficiency, the traditional genetic clinic-based practice has become untenable. Barriers and challenges include low numbers of trained genetic workforce, lack of integrated FHH tools for patients and physicians, and long wait times for available clinic appointments. Further, while cancer syndromes are seen across all groups, gaps in care exist as underserved populations are often not recognized and referred for care.

Investigators propose that these barriers can be overcome by using innovations in informatics and telecommunications to develop a sustainable and scalable genomic care delivery model that can be replicated by other health systems. Such a program would need to integrate FHH applications that collect and analyze family data, SMART-on-FHIR capabilities that can link third party apps with the electronic medical record (EMR), and clinical decision support modules to assist providers and patients. MeTree is one such system with all these capabilities -- a validated and flexible patient-facing FHH collection tool that supports SMART-on-FHIR technology. This platform was the backbone of the Implementing Genomics in Practice (IGNITE) network's FHH clinical utility study that showed clear improvements in the quality and quantity of FHH collected in 5 geographically diverse primary care practices. Furthermore, MeTree was highly acceptable to patients and providers, and was able to properly identify participants at risk for 23 hereditary cancer syndromes for genetic counseling referral.

Our re-submission for this Beau Biden Moonshot grant opportunity is based on the hypothesis that an implementation science approach will improve the identification and management of high-risk patients from diverse clinical setting by systematically integrating FHH driven evidence-based guidelines into the EMR. Investigators plan to improve ascertainment of high-risk patients by imbedding MeTree in the workflow of primary and cancer care clinics. This will improve identification for genetic counseling, facilitate patient education about genetic testing, and risk management for at risk patients, as well as facilitate engagement of patients, family members, and providers with telegenetic and telephone counseling options. This collaborative effort from genetic, genomic, biomedical informatic, and implementation science researchers at Vanderbilt University Medical Center (VUMC), Meharry Medical Center (MMC) and Duke University is highly responsive to the five required elements in RFA-CA-19-017. The proposal has the following specific aims:

SA1. Deploy a care delivery model that will facilitate systematic risk assessment for hereditary cancers in diverse clinical environments.

* 4000 participants will be enrolled and randomized to usual care or MeTree FHH risk assessment
* Deploy in academic medical center (VUMC) and a medical center (MMC) that serves underserved populations
* Assess participants perceptions using online survey and qualitative semi-structured interviews

SA2. Improve access to genetic healthcare providers for participants at risk for hereditary cancer syndromes.

* 300 high risk participants in the VUMC Hereditary Cancer Clinic will be enrolled and randomized
* Extend clinic capacity by lessening the need for in-clinic family history collection and basic counseling
* Expand reach of clinic by using telephone and video genetic counseling, referral to specialists

SA3. Explore the feasibility of our care delivery model to improve family engagement for cancer risk assessment

* Participants extend invitations to MeTree's family resource center to share results of genetic tests
* Assist with education and referral needed for cascade testing for pathogenic variants

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at sites included in study
* Able to read and communicate in English
* Willing to use the Internet
* Currently enrolled in the patient portal, or willing to enroll (VUMC-specific)

Exclusion Criteria:

* Non-study site patient
* Diagnosed with a terminal illness
* Unable to speak/read English
* Unable/unwilling to use the Internet
* Previous genetic testing and/or counseling from the VUMC Hereditary Cancer Clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Anyone over 18 years old, receiving care at our study site (virtual included), and willing/able to use the internet.
Sampling Method: Non-Probability Sample
Enrollment: 1847 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Wiesner, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (2):
- United States (2):
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mittendorf KF, Bland HT, Andujar J, Celaya-Cobbs N, Edwards C, Gerhart M, Hooker G, Hubert M, Jones SH, Marshall DR, Myers RA, Pratap S, Rosenbloom ST, Sadeghpour A, Wu RR, Orlando LA, Wiesner GL. Family history and cancer risk study (FOREST): A clinical trial assessing electronic patient-directed family history input for identifying patients at risk of hereditary cancer. Contemp Clin Trials. 2025 Jan;148:107714. doi: 10.1016/j.cct.2024.107714. Epub 2024 Oct 10. PMID 39395532

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Participants: Participants enrolled in the FOREST observational cohort who were invited to complete study procedures, including a baseline survey and a web-based family health history questionnaire (MeTree). Completion of study components was voluntary, and participants were not assigned to interventions or comparison groups.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 1847
Completed | 620
Not Completed | 1227

BASELINE CHARACTERISTICS:
Population: All participants who were eligible and consented in the study
Groups:
- All Participants: Evaluates the proportion of participants who initiate and complete each step of the FOREST study, including baseline survey and MeTree family health history tool. Data are tracked through REDCap and MeTree backend to measure engagement and completion.
  MeTree Family Health History Tool: A web-based family health history collection and risk assessment platform integrated with EHR systems. Participants complete the MeTree survey, which generates personalized risk reports for hereditary cancer syndromes and provides guideline-based recommendations, including genetic counseling referrals when indicated.
Arm/Group | All Participants
Number analyzed (Participants) | 1847
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1330
  Male | 517
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 1550
  Unknown or Not Reported | 259
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 19
  Native Hawaiian or Other Pacific Islander | 6
  Black or African American | 184
  White | 1435
  More than one race | 0
  Unknown or Not Reported | 197

OUTCOME MEASURES:

1. Primary Outcome: MeTree Completion (REACH)
Description: Proportion of participants sent a MeTree link who complete the MeTree family health history questionnaire, defined by generation of a MeTree risk report. Engagement steps (link clicked, account created) will be summarized descriptively. 95% confidence intervals will be reported using the Wilson method; subgroup comparisons by site and demographics will be exploratory.
Time Frame: From enrollment to study completion (up to 3 years)
Measure: Count of Participants; unit: Participants
Groups:
- Reach: Evaluates the proportion of participants who initiate and complete each step of the FOREST study, including baseline survey and MeTree family health history tool. Data are tracked through REDCap and MeTree backend to measure engagement and completion.
  MeTree Family Health History Tool: A web-based family health history collection and risk assessment platform integrated with EHR systems. Participants complete the MeTree survey, which generates personalized risk reports for hereditary cancer syndromes and provides guideline-based recommendations, including genetic counseling referrals when indicated.
Arm/Group | Reach
Number analyzed (Participants) | 1847
Participants | 1847
Statistical Analysis 1: Comparison: Reach; Paired Pre vs Post MeTree; Test type: Superiority; p < 0.001, McNemar

2. Secondary Outcome: EHR-based Identification for High Risk of Hereditary Cancer (Effectiveness)
Description: Billing code based identification of personal or family history indicators of hereditary cancer
Time Frame: Assessed at two time points: baseline (pre-MeTree, using all available prior EHR history) and 12 months after MeTree completion.
Population: Subset of participants enrolled at VUMC who completed MeTree
Measure: Count of Participants; unit: Participants
Groups:
- EHR-based Identification for High Risk of Hereditary Cancer: We measure the incidence of at-risk designation in our cohort pre- and post-MeTree, using EHR data as a proxy indicator for at-risk status in the pre-MeTree setting (RE-AIM outcome of "Effectiveness").
Arm/Group | EHR-based Identification for High Risk of Hereditary Cancer
Number analyzed (Participants) | 266
Participants
  Pre-MeTree | 155
  Post-MeTree | 111
Statistical Analysis 1: Comparison: EHR-based Identification for High Risk of Hereditary Cancer; Test type: Superiority; p < 0.001, McNemar

3. Secondary Outcome: Genetic Counseling Appointment Lengths
Description: Length of genetic counseling appointments in minutes
Time Frame: At the genetic counseling appointment (index visit) occurring after MeTree results review and within 12 months after enrollment.
Population: Analysis population comprises of 31 MeTree participants who completed MeTree and genetic counseling and 31-non MeTree participants who had genetic counseling appointments at the same clinical over the same time frame as the MeTree study participants
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- MeTree; Standard of Care: Analysis population comprises of 31 MeTree participants who completed MeTree and genetic counseling and 31-non MeTree participants who had genetic counseling appointments at the same clinical over the same time frame as the MeTree study participants
Arm/Group | MeTree | Standard of Care
Number analyzed (Participants) | 31 | 31
Minutes | 45 (15.1) | 48 (15)
Statistical Analysis 1: Comparison: MeTree vs Standard of Care; Test type: Superiority; p = 0.435, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: N/A. Adverse event data was not collected for this study.
Description: No study-related adverse events would reasonably be expected to result from the FOREST study procedures.
Groups:
- All Participants: Participants enrolled in the FOREST prospective observational cohort who were invited to complete study procedures, including a baseline survey and a web-based family health history questionnaire (MeTree). Completion of study components was voluntary. Participants were not assigned to interventions or comparison groups, and results are reported for the overall enrolled population.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/34/NCT05079334/Prot_006.pdf
  • Statistical Analysis Plan (2025-11-03): https://cdn.clinicaltrials.gov/large-docs/34/NCT05079334/SAP_007.pdf
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT05079334/ICF_008.pdf